CLINICAL TRIAL: NCT01905098
Title: Complementary and Alternative Medicine Sauna Detoxification Study: A Phase I Randomized 2-Arm Study to Determine the Impact of Hyperthermia Intervention Protocol on Serum Polychlorinated Biphenyls (PCBs) in Healthy Human Adults.
Brief Title: Complementary and Alternative Medicine Sauna Detoxification Study: Phase I
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bastyr University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: H35B11-Phase1; 5R00AT004711-04 (NIH)
Record Dates: First submitted 2013-07-16; First posted 2013-07-23 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Hyperthermia
Keywords: Detoxification; Sauna; Hyperthermia
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observation-First Arm (Experimental): A group that first attends 4 observation visits without sauna, and then attends sauna sessions 5 times a week for 3.5 hours per visit for 3 weeks.
  Participants in this Arm will undergo both listed interventions: Observation and Sauna Protocols.
  Interventions: Other: Sauna Detoxification Protocol; Other: Observation Sessions
- Sauna-First Arm (Active Comparator): A group that first attends sauna sessions 5 times a week for 3.5 hours per visit for 3 weeks and then attends 4 observation visits without sauna.
  Participants in this Arm will undergo both listed interventions: Observation and Sauna Protocols.
  Interventions: Other: Sauna Detoxification Protocol; Other: Observation Sessions

INTERVENTIONS:
Other: Sauna Detoxification Protocol — All study participants will actively undergo sauna intervention sessions.
  The sauna will be pre-warmed to 160 degrees Fahrenheit and humidity set to 25% +/- 5%. Participants will have a scheduled 10-min break every 30 minutes of sauna, during which time vital signs, symptoms, and fluid intake will be assessed and recorded.
  On a weekly basis, lab assessments will be performed to compare participants' baseline lab values with those during the sauna intervention, and to monitor for safety. In addition, weekly serum samples will be taken for PCB assessment.
  Other Names: Sauna-based detoxification
Other: Observation Sessions — All enrolled participants will undergo observation protocol consisting of one (1) hour visit weekly consistent with Sauna Visits lab assessment time points, to be completed in 3 weeks (4 total sessions within 21 days). At each Observation Visit a blood draw for CBC/D, CMP, and PCBs analysis will be performed, as well as query for symptoms and MOSES questionnaire will be assessed.

SUMMARY:
The purpose of this study is to determine the impact of sauna use on polychlorinated biphenyls (PCB) in the blood of healthy human adults, as well as to assess safety, feasibility, and tolerability, and effects on quality of life and wellness. We hope to determine if there is a link between lower PCB levels in blood and sauna use.

DETAILED DESCRIPTION:
This is a Phase I, 2-Arm randomized trial.

All study participants will actively undergo sauna intervention sessions and observation sessions.

The time between Phone Screen and the End of Study Visit will vary by individual schedule. For the purposes of this study, a participant will be considered 'actively enrolled' when s/he has signed the Full Study Consent Form on the first sauna or observation visit (SV1 or OV1). Each participant will be actively enrolled for at least 7 weeks, but no more than 22 weeks.

All participants will undergo Phone Screen for eligibility prior to participating in any study-related visits. Candidates will first be asked for their oral consent to be screened, and if granted, questioning will continue. If the participant meets pre-screening criteria assessed on the phone, they will be asked to schedule an In-Person Screening Visit.

Prior to randomization, all participants will participate in an In-Person Screening Visit at the Bastyr University (BU) Clinical Research Center (CRC) for: informed consent, to have a blood draw for screening lab analysis, anthropomorphic measurements, a 12-lead ECG assessment, provide demographic data, and medical history assessment.

If participants remain interested and eligible, they will be randomized into either Sauna-First Arm or Observation-First Arm within 2 weeks of eligibility ascertainment using block randomization scheme.

Participants will know that they are in an intervention, but will not know their PCB levels, or the results of questionnaire assessments until approximately three months after the end of the study. The PI will review monitoring and AE data, but will be blinded to PCB data during analysis.

After screening, randomization, and informed consent, study participants in either Arm will either complete a 3-week observation period followed by a 3-week medically monitored sauna-based detoxification intervention; or will first complete a 3-week medically monitored sauna-based detoxification intervention, followed by a 3-week observation period. Each participant will also have an End of Study Visit at least 7 days after the last study visit (Sauna or Observation Visit -depending on the Arm).

The sauna will be pre-warmed to 160 degrees Fahrenheit and humidity set to 25% +/- 5%. Participants will have a scheduled 10-min break every 30 minutes of sauna, during which time vital signs, symptoms, and fluid intake will be assessed and recorded.

During Sauna Visits weekly lab assessments will be performed to compare participants' baseline lab values with those during the sauna intervention, and to monitor for safety. In addition, weekly serum samples will be taken for PCB assessment.

During each Observation Visit a blood draw for Complete Blood Count with Differential (CBC/D), Comprehensive Metabolic Panel (CMP), and PCBs analysis will be performed, as well as query for symptoms and MOSES questionnaire will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 21-35 years.
* Body mass index (BMI) 19 to 29.9 kg/m2 at the screening evaluation.
* Ability to schedule and attend daily visits for the duration of the study.
* If female, willingness to use barrier contraception (e.g., cervical cap, diaphragm, condom, metal (non- hormone) Intrauterine Device (IUD) throughout the study and take a pregnancy test at screening and weekly during the study.

Exclusion Criteria:

* Pregnant, or trying to become pregnant in the three months following screening.
* Current use of any prescribed pharmaceutical medications (including oral contraceptive pills (OCPs) and dietary supplements).
* Refusal to stop taking self-prescribed dietary supplements and OCPs for the duration of the study.
* BMI greater than 29.9 kg/m2 or less than 19 kg/m2.
* Elevated fasting blood sugar (above 125 mg/dL).
* Abnormal ECG findings of: bradycardia (heart rate below 60) not due to athletic bradycardia, ventricular arrhythmias, axis deviation, coronary circulation problems (ischemia/infarct/injury), or any activation sequence disorders (e.g. Right/Left Bundle Branch Block (RBBB/LBBB) and Wolff-Parkinson-White Syndrome (WPW).)
* Hyper or hypotension (BP above 180/100 or below 80/50 respectively).
* A reported diagnosis of any chronic medical condition (e.g., multiple sclerosis, diabetes, or endocrine disorders, liver disease, kidney disease, HIV/AIDS, or cancer), or with a reported history of substance abuse or mental illness within the past 5 years, or a mental health disorder in the past 6 months.
* CBC/D, ALT-Liver Protein, AST-Liver Protein, Blood Urea Nitrogen (BUN), or Creatinine outside of 15% of the Lower/Upper Limit of Normal (LLN/ULN) values.
* Recent infection (<14 days), open sores, or communicable skin conditions.
* Current reported use of any tobacco products or illicit drugs.
* Any condition that, in the opinion of the investigators or Institutional Review Board (IRB), would preclude the safe completion of the study (e.g., clinical or mental health concerns that arise from the overall screening or medical history assessment).
* Previous participation in the pilot sauna detoxification study, and/or participation in a detoxification program within the last 6 months of the Phone Screen.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Impact of sauna protocol on PCB levels | 6 weeks
  The primary comparison measure will be PCB levels at Sauna Visit 15 in the sauna-first Arm and Observation Visit 4 in the Observation-First Arm.
Safety | 6 weeks
  To evaluate the safety of sauna detoxification by recording and describing all adverse events (AE's) throughout the study.

SECONDARY OUTCOMES:
Participant-Reported Symptoms | 6 weeks
  To describe changes in quality of life and participant-reported symptoms associated with participation in the study.
  Query for symptoms will be recorded daily during all sauna visits (SV1-15), at each observation visit (OV1-4), and at the End of Study Visit.
  The RAND Short Form 36 Questionnaire, and NIH Patient-Reported Outcomes Measurement Information System (PROMIS) Questionnaires: Global Wellness, Fatigue, Physical Function will be assessed at SV1, OV1, and End of Study Visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Allen, ND, MPH, Principal Investigator — Bastyr University Research Institute
Locations (1):
- Bastyr University Research Institute, Clinical Research Center, Kenmore, Washington, United States